CLINICAL TRIAL: NCT04000542
Title: Community Pharmacist Use of Mobile ECG to Inform Drug Therapy Decision Making for Patients Receiving QT Prolonging Medications
Brief Title: Pharmacist Use of ECG to Inform Drug Therapy Decisions for Patients Receiving QT Prolonging Medications
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northeast Iowa Medical Education Foundation (Other)
Responsible Party: Principal Investigator, Jim Hoehns, Research Director, Northeast Iowa Medical Education Foundation
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 19-0005
Record Dates: First submitted 2019-06-25; First posted 2019-06-27 (Actual); Last update posted 2020-04-09 (Actual); Status verified 2020-04

CONDITIONS: Torsades de Pointe Caused by Drug (Disorder); Torsades de Pointes; Qt Interval, Variation in
MeSH Terms: conditions — Torsades de Pointes

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Eligible Participants (Experimental): Eligible Participants that consent will receive the pharmacist intervention.
  Interventions: Other: Pharmacist Intervention

INTERVENTIONS:
Other: Pharmacist Intervention — The pharmacist will record a 30 second rhythm strip from patients using the KardiaMobile device and calculate the QTc interval using the Bazett calculation formula. The pharmacist will discuss the result with the patient and if necessary, will contact the prescriber to effect a medication change. If the QTc interval is greater than the 99th percentile, (470 ms for males, 480 ms for females) the pharmacist must contact the prescriber. The pharmacist will record any prescription changes which resulted from the intervention and the prescriber response. The pharmacist will email the rhythm strip (with study participation number) to a secure email at the Northeast Iowa Family Practice Center (NEIFPC). Rhythm strips will be archived for future potential research evaluation in a secure, electronic file.

SUMMARY:
Torsade de pointes (TdP) is a cardiac arrhythmia associated with QT interval prolongation which may lead to cardiac arrest. Prescription medications which cause QT interval prolongation are commonly used in daily practice. To lessen risk of TdP, pharmacists work to minimize combinations of QT interval prolonging drugs. If community pharmacists had real-time information about a patient's QT interval duration, this would have the direct ability to inform their decision making about which patients may be at highest risk of TdP and who may need heightened avoidance of QT prolonging drugs. This project will provide 3 community pharmacies with mobile ECG devices to easily determine QT intervals among patients who have a prescription profile alert for QT interval prolongation. Study outcomes will include: frequency of QT interval prolongation, changes in drug therapy related to QT interval determination, and patient and pharmacist satisfaction with having pharmacist assessment of QT interval.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female at least 18 years of age.
2. Subject is receiving a prescription medication for which there is a "QT/QTc interval prolongation" alert observed on the dispensing pharmacy prescription software.
3. English speaking

Exclusion Criteria:

1. Patients with implantable pacemakers or automatic implantable cardioverter defibrillators
2. Mental condition rendering the subject unable to understand the nature, scope, and possible consequences of the study.
3. Patient has known atrial or ventricular arrhythmia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2019-07-11 (Actual); Primary Completion 2020-03-31 (Actual); Study Completion 2020-03-31 (Actual)

PRIMARY OUTCOMES:
Frequency of medication order changes due to QTc interval prolongation | through study completion (anticipated to last 8 months)
  Physician/provider will be contacted if elevated QTc interval is present (>470 ms for males, >480 ms for females). Frequency of medication changes due to QTc interval prolongation will be assessed.

CONTACTS AND LOCATIONS:
Locations (1):
- Northeast Iowa Family Practice, Waterloo, Iowa, United States

IPD SHARING:
Plan to Share IPD: No